CLINICAL TRIAL: NCT01198158
Title: Randomized Phase III Trial Comparing Everolimus Versus Everolimus Plus Bevacizumab for Advanced Renal Cell Carcinoma Progressing After Treatment With Tyrosine Kinase Inhibitors
Brief Title: Everolimus With or Without Bevacizumab in Treating Patients With Advanced Kidney Cancer That Progressed After First-Line Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-02603; NCI-2011-02603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000684313; CALGB 90802 (Other: Alliance for Clinical Trials in Oncology); CALGB-90802 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Everolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (everolimus) (Active Comparator): Patients receive everolimus PO QD on days 1-28.
  Interventions: Drug: Everolimus; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm II (everolimus with bevacizumab) (Experimental): Patients receive everolimus PO QD on days 1-28 and bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Biological: Bevacizumab; Drug: Everolimus; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm II (everolimus with bevacizumab)
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase III trial studies giving everolimus together with bevacizumab to see how well it works compared to everolimus alone in treating patients with advanced kidney cancer that progressed after first-line therapy. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can interfere with tumor growth by blocking the ability of tumor cells to grow and spread. Everolimus and bevacizumab may also stop the growth of kidney cancer by blocking blood flow to the tumor. It is not yet known whether giving everolimus together with bevacizumab is better than everolimus alone in treating patients with advanced kidney cancer that has progressed after first-line therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To compare the overall survival of patients receiving bevacizumab plus everolimus and everolimus alone among patients with advanced renal cell carcinoma progressing after first line vascular epidermal growth factor receptor (VEGFR)-tyrosine kinase inhibitor (TKI) treatment.

SECONDARY OBJECTIVES:

I. To compare the progression-free survival and proportion who experience an objective response (defined as complete clinical response [cCR] + partial response [PR]) in patients with advanced renal cell carcinoma receiving bevacizumab plus everolimus and everolimus alone.

II. To compare grade 3 or higher toxicity in patients receiving each treatment regimen.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive everolimus orally (PO) once daily (QD) on days 1-28.

ARM II: Patients receive everolimus PO QD on days 1-28 and bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 8 weeks until disease progression and then every 6 months for up to 5.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Renal cell carcinoma with some component of clear cell histology
* Metastatic or unresectable disease
* Must have been treated with at least 1 prior VEGFR tyrosine kinase inhibitor treatment and have progressed or have been intolerant to treatment
* No prior systemic therapy with a vascular endothelial growth factor (VEGF) binding agent (e.g., bevacizumab)
* No prior systemic therapy with any mechanistic target of rapamycin (mTOR) inhibitor (e.g., sirolimus, temsirolimus, everolimus)
* Prior cytokine therapy is allowed
* Any systemic therapy must be completed at least 4 weeks prior to registration
* >= 2 weeks since any prior radiation (including palliative)
* Patients must not have had a major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to study registration, and must have fully recovered from any such procedure

  * The following are not considered to be major procedures: thoracentesis, paracentesis, port placement, laparoscopy, thoracoscopy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies and routine dental procedures
* Patients must have measurable disease by RECIST criteria; lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan
* No active brain metastases: patients with treated, stable brain metastases for at least three months are eligible as long as they meet the following criteria:

  * Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 3 months, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or CT) (stable dose of anticonvulsants are allowed); treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician; patients with central nervous system (CNS) metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 are not eligible
  * Baseline brain imaging (MRI/CT) is required
* No serious non-healing wound, ulcer, or bone fracture
* No arterial thrombotic events within 6 months of registration:

  * Including transient ischemic attack (TIA), cerebrovascular accident (CVA), peripheral arterial thrombus, unstable angina or angina requiring surgical or medical intervention in the past 6 months, or myocardial infarction (MI); patients with clinically significant peripheral artery disease (i.e., claudication on less than one block), significant vascular disease (i.e., aortic aneurysm, history of aortic dissection), or any other arterial thrombotic event are ineligible
* Patients who have experienced a deep venous thrombosis or pulmonary embolus within the past 6 months must be on stable therapeutic anticoagulation to be enrolled to this study
* Patients receiving anti-platelet agents and prophylactic anticoagulation are eligible
* No inadequately controlled hypertension: (defined as a blood pressure of >= 160 mmHg systolic and/or >= 90 mmHg diastolic on medication), or any prior history of hypertensive crisis or hypertensive encephalopathy
* No known severe impairment of lung function, defined as >= grade 2 dyspnea or cough, or either:

  * Requirement of supplemental oxygen, or
  * In cases where pulmonary function or pulse oximetry tests have been obtained, forced expiratory volume of the lung in one second (FEV1) or forced vital capacity (FVC) are < 50% of predicted, or single breath diffusing capacity of the lung for carbon monoxide (DLCO) is < 35% of predicted or resting room oxygen saturation is less than 90%
* No active or severe liver disease (e.g. acute or chronic hepatitis, cirrhosis)
* No positive serology for anti-hemoglobin C (HBC) or anti-hepatitis C virus (HCV) antibodies; hepatitis B virus (HBV) seropositive patients (hepatitis B surface antigen [HBsAg] positive) are eligible if they are closely monitored for evidence of active HBV infection by HBV deoxryribonucleic acid (DNA) testing and agree to receive suppressive therapy with lamivudine or other HBV-suppressive therapy until at least 4 weeks after the last dose of everolimus
* No New York Heart Association (NYHA) class >= 2 congestive heart failure
* No active bleeding or chronic hemorrhagic diathesis or increased risk for bleeding: Including but not limited to history of major bleeding within 6 months (e.g. gastrointestinal, lung, CNS sites; or required transfusion support)
* No history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to the initiation of treatment
* No ongoing immunosuppressive therapy: including chronic systemic treatment with corticosteroids (>= 10 mg/day prednisone equivalent)
* Archival tissue must be available for submission: though it is optional patients to choose to participate in the correlative substudies or not
* Patients who are pregnant or nursing are not eligible

  * Women of child bearing potential must have a negative serum or urine pregnancy test within 16 days prior to registration
  * Women of child-bearing potential include:

    * Any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea >= 12 consecutive months)
    * Women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35m IU/mL
    * Women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy)
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2 or Karnofsky score >= 60%
* Granulocytes >= 1,500/μL
* Platelet count >= 100,000/μL
* Calculated creatinine clearance >= 30 mL/minute (modified Cockroft and Gault formula)
* Bilirubin =< 1.5 x upper limits of normal
* Aspartate aminotransferase (AST) =< 2.5 x upper limits of normal (ULN)
* Fasting serum triglycerides =< 200 mg/dL
* Serum cholesterol =< 300 mg/dL
* Fasting serum glucose =< 1.5 x ULN
* Urine protein to creatinine ratio < 1.0 or urine protein =< 1+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Philips, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (524):
- United States (524):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Providence Medical Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Weill Medical College of Cornell University, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Marion L Shepard Cancer Center at Vidant Beaufort Hospital, Washington, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma-Lakeside, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Mid-Columbia Medical Center/Celilo Cancer Center, The Dalles, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology SC-Appleton, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Everolimus): Patients receive everolimus 10mg daily orally plus intravenous placebo on day 1 and 15 (control arm) in a 28 day cycle.
- Arm II (Everolimus With Bevacizumab): Patients receive everolimus 10mg daily orally plus intravenous bevacizumab 10mg/kg intravenously on day 1 and 15 (experimental arm) in a 28 day cycle.
Period: Overall Study
Arm/Group | Arm I (Everolimus) | Arm II (Everolimus With Bevacizumab)
Started | 41 | 36
Completed | 41 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Everolimus) | Arm II (Everolimus With Bevacizumab) | Total
Number analyzed (Participants) | 41 | 36 | 77
Age, Continuous [Median (Full Range); unit: years] | 62.9 [41.6 to 78.7] | 62 [30.2 to 85.0] | 62.2 [30.2 to 85.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 28 | 31 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 32 | 67
  Non-White | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 36 | 77
Dominant clear cell histology [Count of Participants; unit: Participants] | 34 | 30 | 64

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: The time from date of randomization to date of death due to any cause, assessed up to 5.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Everolimus) | Arm II (Everolimus With Bevacizumab)
Number analyzed (Participants) | 41 | 36
months | 27.5 [14.5 to 34] | 21.8 [14.8 to 27.2]
Statistical Analysis 1: Comparison: Arm I (Everolimus) vs Arm II (Everolimus With Bevacizumab); Test type: Superiority; p = 0.739, Log Rank; OS was analyzed based on an intent-to-treat approach using the stratified log-rank statistic adjusting on the stratification factors

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: The time from randomization to disease progression or death from any cause, assessed up to 5.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Everolimus) | Arm II (Everolimus With Bevacizumab)
Number analyzed (Participants) | 41 | 36
months | 7.2 [3.7 to 9.8] | 6.9 [4.1 to 11.2]
Statistical Analysis 1: Comparison: Arm I (Everolimus) vs Arm II (Everolimus With Bevacizumab); Test type: Superiority; p = 0.832, Log Rank; PFS was analyzed based on an intent-to-treat approach using the stratified log-rank statistic adjusting on the stratification factors

3. Secondary Outcome: Objective Response Rate (CR + PR)
Description: The response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients.
Time Frame: Up to 5.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Everolimus) | Arm II (Everolimus With Bevacizumab)
Number analyzed (Participants) | 41 | 36
percentage of participants | 17.1 [7.2 to 32.1] | 16.7 [6.4 to 32.8]

4. Secondary Outcome: Toxicities, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The number of patients reporting grade 3 or higher adverse events as graded by the NCI's Common Toxicity Criteria (CTCAE) Version 4 are reported here. A complete list of all reported adverse events is reported in the Adverse Events section of this report.
Time Frame: Up to 30 days after completion of study treatment
Population: All patients that started protocol treatment and were assessed for adverse events were included in this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Everolimus) | Arm II (Everolimus With Bevacizumab)
Number analyzed (Participants) | 38 | 33
Participants
  Grade 3 Adverse event | 21 | 20
  Grade 4 Adverse event | 1 | 3

ADVERSE EVENTS:
Time Frame: Up to 30 days after completion of study treatment
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation & scientific analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients with at least 1 cycle of tx and 1 AE form. Serious AE (SAE) reports may include any secondary serious/non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Arm I (Everolimus) | Arm II (Everolimus With Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 33/41 | 28/36
Serious Adverse Events (participants affected / at risk) | 9/38 | 11/33
Other Adverse Events (participants affected / at risk) | 32/38 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Everolimus) (N=38) | Arm II (Everolimus With Bevacizumab) (N=33)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 8 (9)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (7) | 5 (7)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (3)
Cholesterol high (Investigations) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 5 (5) | 6 (9)
INR increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 4 (4)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6) | 4 (7)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3) | 4 (7)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Everolimus) (N=38) | Arm II (Everolimus With Bevacizumab) (N=33)
Anemia (Blood and lymphatic system disorders) | 22 (163) | 21 (116)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (27) | 15 (41)
Mucositis oral (Gastrointestinal disorders) | 11 (16) | 7 (7)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (6)
Edema limbs (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 20 (116) | 23 (92)
Pain (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 3 (4) | 5 (7)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (8) | 4 (7)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (12) | 7 (22)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 17 (92) | 17 (63)
Creatinine increased (Investigations) | 15 (75) | 22 (87)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (13) | 2 (2)
Platelet count decreased (Investigations) | 6 (35) | 13 (31)
Weight loss (Investigations) | 0 (0) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (86) | 21 (90)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 23 (100) | 24 (90)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 4 (13)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 12 (34) | 9 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Hypertension (Vascular disorders) | 10 (74) | 12 (60)
Thromboembolic event (Vascular disorders) | 1 (2) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT01198158/Prot_SAP_000.pdf